CLINICAL TRIAL: NCT04569812
Title: Providing the Best Chest Compression Quality: Standard CPR Versus Chest Compressions Only in a Bystander Resuscitation Model.
Brief Title: Standard CPR Versus Chest Compressions Only
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: St. John's Ambulance, Vienna Austria (Unknown); Universitäres Simulationszentrum Wien, Klinik Floridsdorf, Vienna, Austria (Unknown)
Responsible Party: Principal Investigator, Bernhard Roessler, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1136/2015
Record Dates: First submitted 2019-09-09; First posted 2020-09-30 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: Manikins; Bystander; Quality
MeSH Terms: interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Intervention Model Description: prospective, randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard CPR (Experimental): After Informed Consent Document (ICD) signature, participants were randomised (to the Standard CPR group) to perform standard CPR (30:2) in a flowchart-assisted resuscitation for 5min in a manikin model
  Interventions: Procedure: Cardiopulmonary Resuscitation
- Chest compressions only (Experimental): After ICD signature, participants were randomised (to the CC only CPR group) to perform chest compressions only in a flowchart-assisted resuscitation for 5min in a manikin model
  Interventions: Procedure: Cardiopulmonary Resuscitation

INTERVENTIONS:
Procedure: Cardiopulmonary Resuscitation — flowchart-assisted standard resuscitation or chest compressions-only resuscitation for 5min

SUMMARY:
Background:

More than two thirds of sudden cardiac arrests are witnessed by bystanders. Bystander cardiopulmonary resuscitation (CPR) doubles survival from cardiac arrest. Importantly, even in witnessed cardiac arrests only 20% of the bystanders commence basic life support. Common reasons for not commencing include panicking and the perceived inability to perform CPR correctly. A meta-analysis could demonstrate that a simplification of the algorithm (compression-only dispatcher-assisted bystander CPR) led to a 22% increase in survival-to-hospital discharge. A recently published trial of the research group could demonstrate that the presence of a flowchart has a positive effect on the quality of BLS while at the same time increasing the rescuers' confidence. Nonetheless, performing CPR is exhausting. Previous publications have emphasized increasing fatigue with the duration of CPR efforts in both, standard and chest compressions-only CPR. Consequently, the investigators wanted to test the hypothesis that chest compressions (CC) are delivered more correctly regarding the depth when utilizing the standard Basic Life Support (BLS) algorithm with the aid of a flowchart as compared to the CC only algorithm utilizing an adapted CPR flowchart in a manikin resuscitation model.

Methods:

After consent of the Research Ethics Board of Medical University of Vienna and obtaining written informed consent of the participants, 84 medically untrained laypersons will be randomised to perform flow-chart assisted CPR for 300s following standard CPR guidelines or CC only CPR. The primary outcome parameter will be the total number of CC achieving the correct depth of 50-60mm. Secondary outcome parameters will be hands-off time, the total number of CC, and the compression rate. The total number of delivered rescue breaths, tidal volume, and time to deliver these will also be evaluated. Furthermore, the subjective point of exhaustion affecting the CPR quality, the reason for discontinuation of CPR if stopped within the 300sec. period and the exhaustion at the end of the CPR measures will be evaluated.

DETAILED DESCRIPTION:
Volunteers will be invited to participate in the trial by the study personnel. Recruitment will be conducted at a Training Centre of St. John ambulance, Vienna, Austria, before the starts of the lessons. After giving written informed consent, participants will be randomized using a web based randomization program (www.random.org) and allocated to perform standard CPR or CC only. The randomization for group allocation will be kept in opaque and sealed envelopes.

The evaluation will be performed with an independent investigator using a computer attached Resusci-Anne Skillreporter by Laerdal-Medical® and the Laerdal Skillreporter Software with Segstat (Version 2.3.0, Laerdal Medical, Stavanger, Norway).

The participants will be asked to perform BLS for five minutes on a manikin. The participants will then be asked to undertake any action they deem necessary to rescue the person simulated by the resuscitation manikin. Participants will not be informed about the underlying hypothesis or the outcome parameters. The room will be prepared to minimise outside interruptions.

Additionally, participants will be instructed to indicate the point in time during CPR when they feel that their fatigue is affecting the quality of the life support performed. ("During CPR and without stopping your actions, please tell us "NOW" when you perceive your fatigue is affecting the quality of the life support performed.)

Participants in both groups will receive one of the charts right at the beginning of the scenario with the information that "this chart will provide information on how to perform CPR" and with the start of the clock further instructions regarding is content. Both groups will not receive any further introduction or support. At the beginning of the scenario, the manikin will be positioned in a supine position on the floor. There will be no clock visible for the participant while performing CPR. An investigator is acting as bystander able to call the emergency medical service or to be sent to look for an automated external defibrillator (which will not be available in the scenario). Nonetheless, the investigator is instructed not to provide any information on how to perform CPR and does not physically take part in the primary check, CC, or mouth-to-mouth ventilations.

Data of steps performed or left out will be documented in hardcopy on the case report form by an investigator and the exact times and details of chest compressions and ventilations will be documented electronically (Laerdal Skillreporter Software with Segstat (Version 2.3.0, Laerdal Medical, Stavanger, Norway)). Checklists of necessary steps will be created based on the European Resuscitation Council (ERC) BLS Guidelines 2010 in the same manner as published previously [Roessler et al. 2007, Koster et al. 2010].

After the five-minute period has ended, the participants will be informed that the emergency medical service is now taking over and that they can stop performing CPR. Directly thereafter, they will be asked the following questions "How exhausted are you now on a scale from 1 to 10, where 1 indicates no exhaustion at all and 10 maximum exhaustion?" (Lickert Like 1-10). If a participant chooses to abort resuscitation attempts before the five minutes are over, the open-ended question "Why did you discontinue the resuscitation attempts?" will be raised.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of non-medical professions

Exclusion Criteria:

* <18years
* medical professionals
* known pregnancy
* physical impairments or illnesses that prohibited physical

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2016-04-20 (Actual); Study Completion 2016-04-20 (Actual)

PRIMARY OUTCOMES:
total number of CCs that achieved the correct depth of 5-6cm | During 5 minutes CPR
  correct compression depth according to ERC Guideline 2015

SECONDARY OUTCOMES:
hand-off time | During 5 minutes CPR
  defined as the sum of the total time in which no CCs were provided
time to the administration of CCs | During 5 minutes CPR
  Interval from cardiac arrest to start of chest compressions
total number of CCs | During 5 minutes CPR
  Total number of chest compressions delivered
relative number of correct CCs (%) | During 5 minutes CPR
  Percentage of chest compressions delivered at the correct depth
During 5 minutes CPR | During 5 minute CPR
  chest compressions delivered at a depth of >5cm
relative number of CCs >5cm | During 5 minutes CPR
  percentage of chest compressions delivered at a depth of >5cm
average compression rate | During 5 minutes CPR
  average rate of chest compressions (X/minute)
Time to fatigue | During 5 minutes CPR
  Interval to the timepoint when participants subjectively felt a loss in the quality of CPR due to fatigue
levels of confidence | During 5 minutes CPR
  10-item Likert-like scale
levels of exhaustion | During 5 minutes CPR
  Exhaustion after 5 minutes of CPR (10-item Likert-like scale)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Roessler, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sans S, Kesteloot H, Kromhout D. The burden of cardiovascular diseases mortality in Europe. Task Force of the European Society of Cardiology on Cardiovascular Mortality and Morbidity Statistics in Europe. Eur Heart J. 1997 Dec;18(12):1231-48. No abstract available. PMID 9508543
- [Background] Hasselqvist-Ax I, Riva G, Herlitz J, Rosenqvist M, Hollenberg J, Nordberg P, Ringh M, Jonsson M, Axelsson C, Lindqvist J, Karlsson T, Svensson L. Early cardiopulmonary resuscitation in out-of-hospital cardiac arrest. N Engl J Med. 2015 Jun 11;372(24):2307-15. doi: 10.1056/NEJMoa1405796. PMID 26061835
- [Background] Larsen MP, Eisenberg MS, Cummins RO, Hallstrom AP. Predicting survival from out-of-hospital cardiac arrest: a graphic model. Ann Emerg Med. 1993 Nov;22(11):1652-8. doi: 10.1016/s0196-0644(05)81302-2. PMID 8214853
- [Background] Nolan JP. Cardiac Arrest and Cardiopulmonary Resuscitation. Semin Neurol. 2017 Feb;37(1):5-12. doi: 10.1055/s-0036-1597832. Epub 2017 Feb 1. PMID 28147412
- [Background] Savastano S, Vanni V. Cardiopulmonary resuscitation in real life: the most frequent fears of lay rescuers. Resuscitation. 2011 May;82(5):568-71. doi: 10.1016/j.resuscitation.2010.12.010. Epub 2011 Feb 17. PMID 21333434
- [Background] Perkins GD, Handley AJ, Koster RW, Castren M, Smyth MA, Olasveengen T, Monsieurs KG, Raffay V, Grasner JT, Wenzel V, Ristagno G, Soar J; Adult basic life support and automated external defibrillation section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 2. Adult basic life support and automated external defibrillation. Resuscitation. 2015 Oct;95:81-99. doi: 10.1016/j.resuscitation.2015.07.015. Epub 2015 Oct 15. No abstract available. PMID 26477420
- [Background] Hupfl M, Selig HF, Nagele P. Chest-compression-only versus standard cardiopulmonary resuscitation: a meta-analysis. Lancet. 2010 Nov 6;376(9752):1552-7. doi: 10.1016/S0140-6736(10)61454-7. Epub 2010 Oct 14. PMID 20951422
- [Background] Rossler B, Ziegler M, Hupfl M, Fleischhackl R, Krychtiuk KA, Schebesta K. Can a flowchart improve the quality of bystander cardiopulmonary resuscitation? Resuscitation. 2013 Jul;84(7):982-6. doi: 10.1016/j.resuscitation.2013.01.001. Epub 2013 Jan 7. PMID 23306815